CLINICAL TRIAL: NCT02805387
Title: Bicarbonate, a New Treatment of Labour Dystocia
Brief Title: Bicarbonate Given During Dystocic Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Senior lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Arrested Labor
Keywords: labor dystocia
MeSH Terms: conditions — Dystocia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no treatment (No Intervention): Dystocic women where no bicarbonate was given
- Treatment (Experimental): Dystocic women where bicarbonate was ingested
  Interventions: Dietary Supplement: Treatment

INTERVENTIONS:
Dietary Supplement: Treatment — Bicarbonate was ingested
  Arms: Treatment

SUMMARY:
Dystocic deliveries and the use of bicarbonate

DETAILED DESCRIPTION:
A randomized controlled trial of 200 primiparous women in active labour.If cervical dilation crossed the action line in the partogram or if labour progress was arrested for two hours or more the delivery was considered to be dystocic, and Oxytocin was suggested for stimulation. Inclusion criteria were: primiparity, singleton pregnancy, with an arrested labour progress with a need for oxytocin. Gestational age was between 37-42 weeks, and no maternal /fetal chronic and/or pregnancy-related conditions. Excluded were multiparous women, deliveries with non-cephalic presentation, multiples, deliveries with fetal chronic and/or pregnancy-related conditions, IUFD (Intra Uterine Fetal Death) or premature < 37 weeks of gestation. A randomization into two groups was performed. One group was treated with two bags of Samarin® (=Samarin® group, 5g bicarbonate) one hour before stimulation with oxytocin started. The other group (=nonSamarin® group) received no bicarbonate and started oxytocin immediately, according to local clinical guidelines. Maternal and fetal data was collected from medical files after delivery and analysed according to group.

ELIGIBILITY:
Inclusion Criteria:

* primiparity, singleton pregnancy
* with an arrested labour progress according to the partogram with a need for oxytocin
* Gestational age was between 37-42 weeks
* and no maternal /fetal chronic and/or pregnancy-related conditions.

Exclusion Criteria:

* multiparous women
* deliveries with non-cephalic presentation
* multiples
* deliveries with fetal chronic and/or pregnancy-related conditions
* IUFD (Intra Uterine Fetal Death) or premature < 37 weeks of gestation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Frequency of spontaneous vaginal delivery | during labor

CONTACTS AND LOCATIONS:
Overall Officials: Per Tornvall, professor, Study Chair — Karolinska Institutet
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No